CLINICAL TRIAL: NCT04266210
Title: Clinical Evaluation Two Restorative Systems in Non-carious Cervical Lesions at Patients With Different Systemic Diseases
Brief Title: Clinical Evaluation of a Restorative Glass Ionomer and a Composite Resin for the Restoration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dr. Fatma Dilşad Öz, Assistant Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Glass ionomer - Composite
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Tooth Disease
Keywords: non-caries cervical lesions; glass ionomer; composite resin
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fuji Bulk (Experimental): Glass ionomer (Fuji Bulk, GC, Tokyo Japan)
  Interventions: Device: Fuji Bulk
- G-ænial Posterior (Experimental): Posterior composite resin(G-ænial Posterior, GC, Tokyo Japan)
  Interventions: Device: G-ænial Posterior

INTERVENTIONS:
Device: Fuji Bulk — Restorative system
  Arms: Fuji Bulk
Device: G-ænial Posterior — Restorative system
  Arms: G-ænial Posterior

SUMMARY:
The clinical performances of a restorative glass ionomer and a composite resin will be compared in the restoration of non-carious cervical lesions (NCCLs) at patients with systemic diseases.

After recruiting participants with at least 2 NCCLs and at least one systemic disease, all restorations will be placed by a single clinician. All lesions will be cleaned before restoring.

NCCLs will be divided into two groups: a conventional restorative glass ionomer cement [Fuji Bulk (GC, Tokyo Japan) (FB)] and a posterior composite resin [G-ænial Posterior (GC, Tokyo Japan) (GP)] All restorative procedures will be conducted according to manufacturers' instructions. Restorations will be scored using modified United States Public Health Service (USPHS) criteria after a week (baseline) 6, 12, 24, 36 and 48 months. Descriptive statistics will be performed using chi-square tests.

ELIGIBILITY:
Inclusion Criteria:

Patients with at least one systemic disease such as hypertension, cancer in remission after chemotherapy or radiotherapy, diabetes mellitus, hemophilia, heart disease, coronary artery disease, rheumatoid arthritis, chronic obstructive pulmonary disease, lupus eritematozus.

Patients using medications for hypertension, diabetes mellitus, hemophilia, heart disease, coronary artery disease, rheumatoid arthritis, chronic obstructive pulmonary disease, lupus eritematozus.

Patients who are able to attend recall appointments.

Age greater than 18 years who had at least one systemic disease At least two NCCLs needed to be restored.

At least 20 teeth in occlusion.

Exclusion Criteria:

Non-vital teeth

Mobility of teeth

Severe periodontal disease

Heavy bruxism habit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical performances of different restoratiove systems | two years
  Two year results according to USPHS criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)